CLINICAL TRIAL: NCT03194880
Title: Performance Characteristics of AlereCOMBO and Alere q Detect in an HIV PrEP Program in Thailand
Brief Title: Alere COMBO and Alere q Detect in an HIV PrEP Program in Thailand
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Alere, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Alere COMBO & Alere q Detect
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-04

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV testing: At each visit, the DIC HIV testing algorithm will be performed, and additionally, HIV testing by the Anonymous Clinic Algorithm, the Alere™ HIV Combo and the Alere™ q HIV-1/2 Detect. The latter two tests will be performed at the DICs. In case of an invalid result for the Alere™ HIV Combo or the Alere™ q HIV-1/2 Detect, the test will be repeated. If the repeated test is invalid after the second attempt, it is recorded as 'invalid result'.
  Interventions: Device: AlereCOMBO and Alere q Detect

INTERVENTIONS:
Device: AlereCOMBO and Alere q Detect — The feasibility assessment will comprise of two components:
  1. User's perspective: A questionnaire will be developed and used to assess the level of satisfaction among community health workers performing the two new tests, using a 5 point Likert scale. We will assess the training and manual, the use of the test, the user's confidence, troubleshooting and technical support components and resolving problems.
  2. The laboratory component: For each test we will evaluate:
     * The percentage of assays completed
     * The percentage of assays incomplete (i.e. invalid result on two attempts)
     * Reasons for incomplete assays, e.g.
       * The sample could not be delivered to the strip or cartridge correctly
       * Invalid control
       * Results could not be interpreted
       * Others

SUMMARY:
Two new rapid HIV tests by Alere™ have the potential to substantially decrease the window period for rapid tests. First, the Alere™ HIV Combo is a rapid fourth generation test. The performance in a laboratory based setting was recently assessed at the Thai Red Cross Anonymous Clinic Laboratory in Bangkok, Thailand (personal communication). Of 50 confirmed acute HIV samples, Alere™ HIV Combo could detect 37 (74%), while none of these 50 cases could be identified by the currently used third generation tests. These data have not yet been published, but the preliminary results indicate a very favorable performance of the Alere™ HIV Combo in a facility-based laboratory setting.

Second, the Alere™ q HIV-1/2 Detect is a qualitative, cartridge based, nucleic acid amplification test designed for Point of Care use. Data from several early infant diagnosis studies in Sub-Saharan African countries have assessed the performance of the Alere™ q HIV-1/2 Detect. The test was performed in the field, by a range of health professionals, from nurses and laboratory technicians to medical doctors. The pooled analysis showed a sensitivity of 99.07% (95%CI 95.48 - 99.95%) and a specificity of 99.94% (99.72-100%).

DETAILED DESCRIPTION:
This will be a prospective study, collecting blood samples from individuals receiving PrEP at one of two drop-in centers in Bangkok, Thailand:

Rainbow Sky Association of Thailand (RSAT) and Service Worker IN Group (SWING). RSAT is a community-based organization for people with sexual diversity (MSM, gay, transgender, lesbians, and bisexual), and has specific programs for MSM, transgender and lesbian health. SWING promotes HIV prevention among male and female sex workers and provides both community outreach and clinical services at their center. Both locations offer PrEP as part of their service.

Participants who visit the DICs seeking to receive PrEP will undergo HIV testing at several time points: before receiving PrEP (Month 0), one month after starting PrEP (Month 1), three months after starting PrEP (Month 3), and every three months thereafter.

The routine HIV testing algorithm in the DIC is as follows:

* Determine® HIV-1/2 (Alere Medical Co., Ltd.), if reactive followed by two other rapid 3rd generation immunochromatography anti-HIV tests. These are all rapid tests on whole blood as collected by finger prick, performed by trained community health workers in the DIC.

For the purpose of this study, two additional blood samples will be taken by phlebotomy to perform:

* The Anonymous Clinic HIV-testing algorithm (see Annex 1): Architect® HIV-1/2 Combo (Abbott), if reactive followed by Determine® HIV-1/2 (Alere) and Elecsys® HIV combi PT (Roche). Samples that are non-reactive by Architect® HIV-1/2 Combo will be tested by pooled NAAT using Aptima HIV-1 RNA qualitative assay (Hologic®) to screen for acute HIV infection. Samples that are positive by Architect®, Determine® and Elecsys® will be tested by second generation EIA (which detects IgG Ab) to identify acute HIV infection (i.e. 4th generation reactive and 2nd generation negative). This is the standard HIV testing algorithm performed at the Thai Red Cross Anonymous Clinic Laboratory and will identify acute HIV infections.
* Alere™ HIV Combo Alere™ q HIV-1/2 Detect Both the regular DIC algorithm and the Anonymous Clinic algorithm will be used as comparator methods.

ELIGIBILITY:
Inclusion Criteria:

* Will start receiving PrEP at one of the participating clinics
* 18 years or older
* Willing to provide informed consent

Exclusion Criteria:

* Not receiving PrEP at one of the participating clinics
* HIV-infected

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants visiting either the RSAT or SWING drop in centers in Bangkok to access PrEP will be asked to join the study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
HIV test results | 5 years
  The HIV test results will be reported by number and proportions for Alere™ HIV Combo, Alere™ q HIV-1/2 Detect and the standard HIV testing algorithms; the number of acute HIV infections detected by Alere™ HIV Combo and Alere™ q HIV-1/2 Detect will be calculated as the proportion of the total number of participants who have confirmed acute HIV infection. The reliability and validity assessment of Alere™ HIV Combo and Alere™ q HIV-1/2 Detect will be compared with the standard HIV testing and we will present the results as the sensitivity, specificity, number of false positives and number of false negatives. The measuring agreement of HIV test results will be compared between the standard HIV testing algorithms and Alere™ HIV Combo, the standard HIV testing algorithms and Alere™ q HIV-1/2 Detect.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (2):
- Thailand (2):
  - Service Worker IN Group (SWING), Bang Rak, Bangkok
  - Rainbow Sky Association of Thailand (RSAT), Bangkok